CLINICAL TRIAL: NCT06443294
Title: Development of a Smoking Cessation Video Series
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wayne State University (Other)
Responsible Party: Principal Investigator, Michael Schmidt, Graduate Student Researcher, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-23-10-6207
Record Dates: First submitted 2024-04-25; First posted 2024-06-05 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-05

CONDITIONS: Tobacco Use Cessation; Tobacco Smoking
MeSH Terms: conditions — Tobacco Use Cessation; Tobacco Smoking

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video Group (Experimental): Participants randomly assigned to this group will be provided access to the video intervention series.
  Interventions: Behavioral: Smoking cessation video series.
- No-Video Group (No Intervention)

INTERVENTIONS:
Behavioral: Smoking cessation video series. — The intervention in this study is a series of six videos totally approximately 40 minutes. These videos are led by a doctoral psychology student with experience in working with tobacco smokers. Videos utilize empirically-supported strategies for smoking cessation.
  Arms: Video Group

SUMMARY:
This study seeks to develop and test an internet video series aimed at helping individuals reduce cigarette smoking. Participants (daily smokers) will be asked to watch a series of six videos (approximately 6.5 minutes each) which cover various empirically-supported smoking cessation strategies and tools. Examples of strategies included in the videos include noticing smoking cues and consequences and relaxation training. Participants' demographic information, motivation to change, reactions to the video series alliance with video therapist, and confidence in avoiding smoking will all be measured. Additionally, participants will be asked to report their smoking behavior at study baseline and follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Daily smoker
* Interested in reducing smoking
* Not currently enrolled in any smoking cessation program.

Exclusion Criteria:

* Not interested in reducing smoking
* Currently enrolled in a smoking cessation program.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-04-25 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Smoking Quantity/Frequency | Measured at baseline and 30 days following completion of video series.
  Cigarettes smoked in past 30 days.
Subjective Reactions to Video Series | Measured upon completion of video series, within 2 weeks of beginning study.
  Scale based on measure previously developed and used by PI of this study (Schmidt et al., 2023). Outcome explores participants' experience with and opinions of video intervention (e.g., video helpfulness, clarity, etc.).
Self-Efficacy Questionnaire | Measured upon completion of video series (within 2 weeks of beginning study) and at 30-day follow-up.
  Participants' belief in their ability to avoid smoking. SEQ-12: Etter et al., 2000)

SECONDARY OUTCOMES:
The Working Alliance Inventory for Guided Internet Interventions | Measured upon completion of video series, within 2 weeks of beginning study.
  Participants' sense of alliance with therapist leading video intervention. (WAI-I: Penedo et al., 2020).
Motivation to Quit Smoking (Change Ladder) | Measured upon completion of video series (within 2 weeks of beginning study) and one-month follow-up.
  Participants' level of motivation to change smoking behavior measured using a stages of change ladder based in Motivational Interviewing principles.
Smoking Quit Attempt | Measured at 30-day follow-up.
  Whether participants made a quit attempt during the course of the study. Measured using a single, "yes or no" item asking whether participants attempted to quit smoking in the past month.

CONTACTS AND LOCATIONS:
Locations (1):
- Wayne State University, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data is not planned to be shared with other researchers.

REFERENCES:
- [Background] Abroms LC, Lee Westmaas J, Bontemps-Jones J, Ramani R, Mellerson J. A content analysis of popular smartphone apps for smoking cessation. Am J Prev Med. 2013 Dec;45(6):732-6. doi: 10.1016/j.amepre.2013.07.008. PMID 24237915
- [Background] Burman A, Haeder SF, Xu WY. Provider directory inaccuracy and timely access for mental health care. Am J Manag Care. 2023 Feb;29(2):96-102. doi: 10.37765/ajmc.2023.89318. PMID 36811984
- [Background] Grant S, Colaiaco B, Motala A, Shanman R, Booth M, Sorbero M, Hempel S. Mindfulness-based Relapse Prevention for Substance Use Disorders: A Systematic Review and Meta-analysis. J Addict Med. 2017 Sep/Oct;11(5):386-396. doi: 10.1097/ADM.0000000000000338. PMID 28727663
- [Background] Guo YQ, Chen Y, Dabbs AD, Wu Y. The Effectiveness of Smartphone App-Based Interventions for Assisting Smoking Cessation: Systematic Review and Meta-analysis. J Med Internet Res. 2023 Apr 20;25:e43242. doi: 10.2196/43242. PMID 37079352
- [Background] Lee EB, An W, Levin ME, Twohig MP. An initial meta-analysis of Acceptance and Commitment Therapy for treating substance use disorders. Drug Alcohol Depend. 2015 Oct 1;155:1-7. doi: 10.1016/j.drugalcdep.2015.08.004. Epub 2015 Aug 13. PMID 26298552
- [Background] Magill M, Ray L, Kiluk B, Hoadley A, Bernstein M, Tonigan JS, Carroll K. A meta-analysis of cognitive-behavioral therapy for alcohol or other drug use disorders: Treatment efficacy by contrast condition. J Consult Clin Psychol. 2019 Dec;87(12):1093-1105. doi: 10.1037/ccp0000447. Epub 2019 Oct 10. PMID 31599606
- [Background] Richardson CG, Vettese L, Sussman S, Small SP, Selby P. An investigation of smoking cessation video content on YouTube. Subst Use Misuse. 2011;46(7):893-7. doi: 10.3109/10826084.2011.570628. PMID 21599505